CLINICAL TRIAL: NCT06985667
Title: The Effect of the 'Cognitive-Based Behavior Change Training Program' Applied to Parents of Preschool Children With Behavior Problems on Parents' Attitudes and Stress Levels Towards the Child and on the Problematic Behaviors of the Children
Brief Title: Cognitive-Based Behavior Change Training Program
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Uskudar University (Other)
Responsible Party: Principal Investigator, SELMA HASANOĞLU, Principal Investigator, Uskudar University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: E-97105791-050.04-51964
Record Dates: First submitted 2025-04-27; First posted 2025-05-22 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: Behavioral Symptom; Preschool Child; Parent; Parent-Child Relations; Cognitive Ability, General
MeSH Terms: conditions — Behavioral Symptoms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): Implementation of the 8-session parent study
  Interventions: Behavioral: Cognitive-Based Behavior Change Training Program
- Control groups (No Intervention): Group where parental work was not implemented

INTERVENTIONS:
Behavioral: Cognitive-Based Behavior Change Training Program — Parents will be given an 8-session parent training program.
  Session 1: Establishing a trusting relationship and informing them about the study Session 2: Informing parents about the cognitive development of 3-6 year old children Theme: Children learn with 'numbers/scales/amounts' Session 3: Parents being consistent in their approach to children Theme: Children learn with the all/or nothing rule Session 4: Reinforcing positive behaviors in children Theme: Children Learn Laterally Session 5: Parents being positive models Theme: Children Learn by Imitation Session 6: Guidance of parents on the principle of 'learning by doing and experiencing' Theme: Children Learn by Action Session 7: This is the last session. Session 8: Application of final tests and saying goodbye.
  Arms: Experimental Group

SUMMARY:
This study will be conducted to determine the effects of the Parent Education Program Based on the Cognitive Development of the Child, which is applied to the parents of preschool children with behavioral problems, on the attitudes and stress levels of the parents and the problematic behaviors of the children.

The purpose of this study has two dimensions;

Dimension 1: The 'Parent Education Program Based on the Cognitive Development of the Child', which is planned to be developed for the purpose of measuring the attitudes, stress levels of the parents and the effects on the problematic behaviors of the children.

The development of the program was based on Jean Piaget's theory of cognitive development.

Dimension: It is experimental. The aim is to reveal the effectiveness of the Parent Education Program, which will be applied to the parents of children with behavioral problems. There are parent training programs developed for children with behavioral problems in the preschool period. However, the lack of parent studies based on the child's cognitive development reveals the rationale and importance of this study.

ELIGIBILITY:
Inclusion Criteria:

* Children must be between the ages of 3-6
* Participating in the study as a mother and father together
* Not having attended any parent training

Exclusion Criteria:

* Participating in the study as a single parent
* The child must have been diagnosed in the special needs category

Ages: 3 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 44 (Actual)
Dates: Start 2025-04-01 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Preschool Behavior Problems Screening Scale | One month prior to the intervention / One month following the intervention
  The "Preschool Behavior Questionnaire" developed by Behar (1976; Cited in Kanlıkılıçer, 2005) is a Likert-type scale used to determine the behavioral problems of preschool children. The scale was adapted to Turkish by Kanlıkılıçer, and the propositions in the scale were converted into questions and used. The original Turkish version of the "Preschool Behavior Problems Screening Scale" consists of 30 items. After the factor analysis conducted for this study, items with item loading values below .50 were removed, so 15 items were used. The highest score a child can get from the "Preschool Behavior Problems Screening Scale" is "30", and the lowest score is "0".
Parent Stress Scale | One month prior to the intervention / One month following the intervention
  The "Parenting Stress Scale" was developed to measure the stress experienced by parents of children with normal developmental characteristics regarding parenting. The scale consists of 18 items and has a single-dimensional structure that includes the parent, parent-child relationship, and the characteristics of the child. The Parenting Stress Scale is a Likert-type measurement tool evaluated from 0 (Does not describe at all) to 4 (Describes very well). The range of scores that can be obtained from the scale is between 0-72, with higher scores indicating the level of parenting stress. The scale is a measurement tool that can be easily applied to parents with at least one child with a primary school education level or higher.
Parent Attitude Scale | One month prior to the intervention / One month following the intervention
  The Parental Attitude Scale was developed by Evren Karabulut Demir to measure the attitudes of parents with children aged 2 to 6 years, and its validity and reliability study was conducted in collaboration with Gül Erdil. The scale is designed to be applied to parents of children within this age range and consists of 46 items grouped under four subdimensions: Democratic, Authoritarian, Overprotective, and Permissive. The scale is structured in a 5-point Likert format, with each item offering five response options that vary based on frequency or degree of agreement. Participants are asked to indicate their level of agreement with each statement using the following options:
  1 = Strongly disagree, 2 = Disagree, 3 = Neutral, 4 = Agree, and 5 = Strongly agree.
  This Likert-type rating system allows for a quantitative evaluation of parental attitudes across the specified subdimensions. Some items are negatively worded and are therefore reverse-coded prior to analysis. Higher scores within ea

CONTACTS AND LOCATIONS:
Locations (1):
- Gaziantep Municipality Kindergartens, Gaziantep, Gaziantep, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No